CLINICAL TRIAL: NCT02088203
Title: Evaluation of Soy-protein Russian Tarragon (Artemisia Dracunculus L.) Complex as a Dietary Supplement to Improve Carbohydrate Metabolism; Dosing, Safety and Tolerability
Brief Title: Evaluation of Soy-protein Russian Tarragon (Artemisia Dracunculus L.)
Acronym: RT2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); Office of Dietary Supplements (ODS) (NIH)
Responsible Party: Principal Investigator, Jennifer C. Rood, Principal Investigator, Pennington Biomedical Research Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: PBRC 2013-049; P50AT002776 (NIH)
Record Dates: First submitted 2014-02-28; First posted 2014-03-14 (Estimated); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Diabetes Prevention

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (18):
- Single Dose Sequence 1 (Experimental): Dose 1, Dose 2, Dose 0: Each subject will receive a single dose during each of three separate test periods.
  Interventions: Dietary Supplement: Dose 1; Dietary Supplement: Dose 2; Dietary Supplement: Dose 0
- Single Dose Sequence 2 (Experimental): Dose 1, Dose 0, Dose 2: Each subject will receive a single dose during each of three separate test periods.
  Interventions: Dietary Supplement: Dose 1; Dietary Supplement: Dose 2; Dietary Supplement: Dose 0
- Single Dose Sequence 3 (Experimental): Dose 0, Dose 1, Dose 2: Each subject will receive a single dose during each of three separate test periods.
  Interventions: Dietary Supplement: Dose 1; Dietary Supplement: Dose 2; Dietary Supplement: Dose 0
- Single Dose Sequence 4 (Experimental): Dose 3, Dose 4, Dose 0: Each subject will receive a single dose during each of three separate test periods.
  Interventions: Dietary Supplement: Dose 0; Dietary Supplement: Dose 3; Dietary Supplement: Dose 4
- Single Dose Sequence 5 (Experimental): Dose 3, Dose 0, Dose 4: Each subject will receive a single dose during each of three separate test periods.
  Interventions: Dietary Supplement: Dose 0; Dietary Supplement: Dose 3; Dietary Supplement: Dose 4
- Single Dose Sequence 6 (Experimental): Dose 0, Dose 3, Dose 4: Each subject will receive a single dose during each of three separate test periods.
  Interventions: Dietary Supplement: Dose 0; Dietary Supplement: Dose 3; Dietary Supplement: Dose 4
- Single Dose Sequence 7 (Experimental): Dose 5, Dose 6, Dose 0: Each subject will receive a single dose during each of three separate test periods.
  Interventions: Dietary Supplement: Dose 0; Dietary Supplement: Dose 5; Dietary Supplement: Dose 6
- Single Dose Sequence 8 (Experimental): Dose 5, Dose 0, Dose 6: Each subject will receive a single dose during each of three separate test periods.
  Interventions: Dietary Supplement: Dose 0; Dietary Supplement: Dose 5; Dietary Supplement: Dose 6
- Single Dose Sequence 9 (Experimental): Dose 0, Dose 5, Dose 6: Each subject will receive a single dose during each of three separate test periods.
  Interventions: Dietary Supplement: Dose 0; Dietary Supplement: Dose 5; Dietary Supplement: Dose 6
- Multiple Dose Sequence 1 (Experimental): Dose 1, Dose 0, Dose 2: Each subject will receive daily doses for 21 consecutive days during each of three separate test periods.
  Interventions: Dietary Supplement: Dose 1; Dietary Supplement: Dose 2; Dietary Supplement: Dose 0
- Multiple Dose Sequence 2 (Experimental): Dose 1, Dose 2, Dose 0: Each subject will receive daily doses for 21 consecutive days during each of three separate test periods.
  Interventions: Dietary Supplement: Dose 1; Dietary Supplement: Dose 2; Dietary Supplement: Dose 0
- Multiple Dose Sequence 3 (Experimental): Dose 0, Dose 1, Dose 2: Each subject will receive daily doses for 21 consecutive days during each of three separate test periods.
  Interventions: Dietary Supplement: Dose 1; Dietary Supplement: Dose 2; Dietary Supplement: Dose 0
- Multiple Dose Sequence 4 (Experimental): Dose 2, Dose 0, Dose 6: Each subject will receive daily doses for 21 consecutive days during each of three separate test periods.
  Interventions: Dietary Supplement: Dose 2; Dietary Supplement: Dose 0; Dietary Supplement: Dose 6
- Multiple Dose Sequence 5 (Experimental): Dose 2, Dose 6, Dose 0: Each subject will receive daily doses for 21 consecutive days during each of three separate test periods.
  Interventions: Dietary Supplement: Dose 2; Dietary Supplement: Dose 0; Dietary Supplement: Dose 6
- Multiple Dose Sequence 6 (Experimental): Dose 0, Dose 2, Dose 6: Each subject will receive daily doses for 21 consecutive days during each of three separate test periods.
  Interventions: Dietary Supplement: Dose 2; Dietary Supplement: Dose 0; Dietary Supplement: Dose 6
- Multiple Dose Sequence 7 (Experimental): Dose 1, Dose 0, Dose 6: Each subject will receive daily doses for 21 consecutive days during each of three separate test periods.
  Interventions: Dietary Supplement: Dose 1; Dietary Supplement: Dose 0; Dietary Supplement: Dose 6
- Multiple Dose Sequence 8 (Experimental): Dose 1, Dose 6, Dose 0: Each subject will receive daily doses for 21 consecutive days during each of three separate test periods.
  Interventions: Dietary Supplement: Dose 1; Dietary Supplement: Dose 0; Dietary Supplement: Dose 6
- Multiple Dose Sequence 9 (Experimental): Dose 0, Dose 1, Dose 6: Each subject will receive daily doses for 21 consecutive days during each of three separate test periods.
  Interventions: Dietary Supplement: Dose 1; Dietary Supplement: Dose 0; Dietary Supplement: Dose 6

INTERVENTIONS:
Dietary Supplement: Dose 1 — Russian Tarragon Nutrasorb 0.3 g
  Arms: Multiple Dose Sequence 1; Multiple Dose Sequence 2; Multiple Dose Sequence 3; Multiple Dose Sequence 7; Multiple Dose Sequence 8; Multiple Dose Sequence 9; Single Dose Sequence 1; Single Dose Sequence 2; Single Dose Sequence 3
Dietary Supplement: Dose 2 — Russian Tarragon Nutrasorb 1 g
  Arms: Multiple Dose Sequence 1; Multiple Dose Sequence 2; Multiple Dose Sequence 3; Multiple Dose Sequence 4; Multiple Dose Sequence 5; Multiple Dose Sequence 6; Single Dose Sequence 1; Single Dose Sequence 2; Single Dose Sequence 3
Dietary Supplement: Dose 0 — Placebo
Dietary Supplement: Dose 3 — Russian Tarragon Nutrasorb 3 g
  Arms: Single Dose Sequence 4; Single Dose Sequence 5; Single Dose Sequence 6
Dietary Supplement: Dose 4 — Russian Tarragon Nutrasorb 10 g
  Arms: Single Dose Sequence 4; Single Dose Sequence 5; Single Dose Sequence 6
Dietary Supplement: Dose 5 — Russian Tarragon Nutrasorb 20 g
  Arms: Single Dose Sequence 7; Single Dose Sequence 8; Single Dose Sequence 9
Dietary Supplement: Dose 6 — Russian Tarragon Nutrasorb 30 g
  Arms: Multiple Dose Sequence 4; Multiple Dose Sequence 5; Multiple Dose Sequence 6; Multiple Dose Sequence 7; Multiple Dose Sequence 8; Multiple Dose Sequence 9; Single Dose Sequence 7; Single Dose Sequence 8; Single Dose Sequence 9

SUMMARY:
Safety and tolerability of a soy-protein Russian Tarragon complex versus a placebo.

DETAILED DESCRIPTION:
Plants from the genus Artemisia, and specifically Artemisia dracunculus L. (Russian tarragon) have had a long history of medicinal (health) and culinary (food) use and have been reported as effective as a traditional treatments for diabetes in various parts of the world. The overall objective of this study is to conduct early human investigation and to evaluate the effect of nutritional supplementation with a well characterized extract of Artemisia dracunculus L. The primary objectives would be to evaluate safety, tolerability and effective dose in non-diabetic human subjects. Secondary objectives would assess metabolism of the extract and evaluate effects on proposed mechanisms such as insulin secretion, lipid levels and/or insulin resistance.

Single Oral Dose Evaluation

After completing a screening visit and meeting qualifications for the single oral dose evaluation, subjects will receive three single doses (two different doses of the supplement and one dose of placebo) on three separate test periods which are separated by a washout period of at least 7 days. Each testing period requires an overnight stay on the inpatient unit. The inpatient stay will be approximately 26 hours. The doses that will be used in the study are 0.3, 1, 3, 10, 20 and 30 grams plus the placebo. The supplement and the placebo will be mixed with sugar-free flavoring in water. There will be an opportunity to sample the liquid drink during the screening visit.

Screening Visit 1 (about 1 hour) - Fasting (Nothing to eat or drink other than water for at least 10 hours prior to appointment)

* Sign informed consent if willing to participate
* Body weight and height will be measured (body mass index will be calculated from these measures)
* Blood pressure, pulse and temperature will be measured
* Physical exam and ECG (electrocardiogram)
* Report any medications taken over the past 3 months
* Blood draw (about 2 teaspoons) to assess overall health
* Taste test

ALL PROCEDURES AND VISITS LISTED BELOW WILL BE REPEATED 3 TIMES. ALL TESTING WILL BE DONE FOR EACH SINGLE DOSE TESTING PERIOD (1,2,3)

* Testing Period 1: Day -3, Day 1, Day 2
* 7 Day Washout
* Testing Period 2: Day -3, Day 1, Day 2
* 7 Day Washout
* Testing Period 3: Day -3, Day 1, Day 2

Day -3 (about 4 hours) Fasting (Nothing to eat or drink other than water for at least 10 hours prior to appointment)

* Blood pressure, pulse and temperature will be measured
* An IV line will be placed in an arm vein for blood draw purposes and will remain there throughout the testing.
* A blood draw (approximately 2 teaspoons) will be done before and after dosing to assess any changes in glucose or insulin.
* An Oral Glucose Tolerance Test (OGTT) will be done A blood sample will be drawn from the IV line, and then the subject will drink a sugar solution consisting of 75 grams of glucose. Blood will be drawn at specific times after the drink is consumed. Each blood sample will be about 1 tablespoon. (6 tablespoons total for the test). During the IV procedure, a small amount of the subject's own blood (less than 1 teaspoon) will immediately be returned into the vein through the IV after each specimen is collected.
* Adverse events and changes in medication will be assessed by the staff
* Meet with staff briefly about dietary intake and weight maintenance diets

Day 1 (Inpatient Stay- 26 hours) Fasting (Nothing to eat or drink other than water for at least 10 hours prior to appointment)

* Admission to the inpatient unit in the morning of the Day 1 visit. The subject will remain on the unit overnight and be discharged on Day 2.
* Blood pressure, pulse and temperature will be measured.
* Randomization to the study dosing scheme will occur. Randomization is like flipping a coin. The subject and the study staff will not know what dose the subject is receiving or if the subject is receiving a placebo (inactive drink).
* Single dose of extract given (either the supplement or placebo). The dose will be given 2 hours prior to the start of the OGTT. The extract will be in a powder form and will be mixed with up to 8 ounces of liquid for the subject to drink.
* An IV line will be placed in the arm vein for blood draw purposes and will remain there throughout the testing.
* OGTT as described above (at day -3).
* A blood draw (approximately 2 teaspoons) before and after dosing will be done to assess any changes in glucose or insulin. Blood draws will occur at 30, 60, 90, 120, 180, 240 minutes and 12 hours after dosing.
* An ECG will be performed.
* Adverse events and changes in medication will be assessed by the staff.
* The subject will be asked to fast overnight until your blood work on Day 2.

Day 2 (Inpatient) Blood pressure, weight, pulse and temperature will be measured.

* A physical exam will be done
* A 24 hour post dose blood draw (approximately 1 teaspoon) will be done.
* Study staff will schedule the next testing period if applicable and then the subject will be discharged from the inpatient unit.

Multiple Oral Dose Evaluation

After completing a screening visit and meeting qualifications for the multiple oral dose evaluation, subjects will receive three doses (two different doses of the supplement and one dose of placebo) over three separate 21-day test periods that are each separated by a washout period of at least 7 days. Each testing period involves 8 clinic visits. The doses that will be used in the study are 0.3, 1, and 30 grams plus the placebo. The supplement and the placebo will be mixed with sugar-free flavoring in water. There will be an opportunity to sample the liquid drink during the screening visit.

Screening Visit 1 (about 1 hour) - Fasting (Nothing to eat or drink other than water for at least 10 hours prior to appointment)

* Sign informed consent if willing to participate
* Body weight and height will be measured (body mass index will be calculated from these measures)
* Blood pressure, pulse and temperature will be measured
* Physical exam and ECG (electrocardiogram)
* Report any medications taken over the past 3 months
* Blood draw (about 2 teaspoons) and urine collection to assess overall health
* Meet with dietitian about normal dietary intake
* Taste test

ALL PROCEDURES AND VISITS LISTED BELOW WILL BE REPEATED 3 TIMES. ALL TESTING WILL BE DONE FOR EACH MULTIPLE DOSE TESTING PERIOD (1,2,3)

* Testing Period 1: Day -3, Day 1, Day 3, Day 7, Day 10, Day 14, Day 17, Day 21
* 7 Day Washout
* Testing Period 2: Day -3, Day 1, Day 3, Day 7, Day 10, Day 14, Day 17, Day 21
* 7 Day Washout
* Testing Period 3: Day -3, Day 1, Day 3, Day 7, Day 10, Day 14, Day 17, Day 21

Day -3 (about 4 hours) Fasting (Nothing to eat or drink other than water for at least 10 hours prior to appointment)

* Blood pressure, pulse, weight, and temperature will be measured
* An IV line will be placed in an arm vein for blood draw purposes and will remain there throughout the testing.
* An Oral Glucose Tolerance Test (OGTT) will be done. A blood sample will be drawn from the IV line, and then the subject will drink a sugar solution consisting of 75 grams of glucose. Blood will be drawn at specific times after the drink is consumed. Each blood sample will be about 1 tablespoon (3 tablespoons total for the test). During the IV procedure, a small amount of the subject's own blood (less than 1 teaspoon) will immediately be returned into the vein through the IV after each specimen is collected.
* Females of child-bearing potential will have a urine pregnancy test
* A dual-energy X-ray absorptiometry (DXA) scan will be performed using a whole-body scanner. This scan measures the amount of bone, muscle, and fat in the body. The subject will wear a hospital gown, remove all metal-containing objects, and lie down on a table with legs held together by Velcro straps. A scanner emitting low-energy X rays and a detector will pass along the body. The subject is asked to remain completely still for the duration of the 10-minute scan.
* Adverse events and changes in medication will be assessed by the staff
* Meet with staff to assess dietary intake since prior visit

Day 1 (about 45 minutes) Non-fasting

* Blood pressure, pulse, weight, and temperature will be measured.
* Randomization to the study dosing scheme will occur. Randomization is like flipping a coin. The subject and the study staff will not know what dose the subject is receiving or if the subject is receiving a placebo (inactive drink).
* The first dose of extract will be given (either the supplement or placebo). The subject will be given instructions on how to take the extract at home. The extract will be in a powder form to be mixed with up to 8 ounces of liquid to drink.
* Adverse events and changes in medication will be assessed by the staff.

Days 3, 10, and 17 (about 30 minutes each) Non-fasting

* Blood pressure, pulse, weight, and temperature will be measured.
* Compliance with extract dosing will be assessed and additional extract dispensed as needed.
* Adverse events and changes in medication will be assessed by the staff.

Days 7, 14, and 21 (about 6 hours each) Fasting (Nothing to eat or drink other than water for at least 10 hours prior to appointment)

* Blood pressure, pulse, weight, and temperature will be measured.
* Compliance with extract dosing will be assessed and additional extract dispensed as needed (except at Day 21 when dosage is stopped).
* Adverse events and changes in medication will be assessed by the staff.
* Physical exam and ECG (electrocardiogram) will be performed.
* An IV line will be placed in the arm vein for blood draw purposes and will remain there throughout the testing.
* OGTT as described above (at Day -3).
* A blood draw (approximately 3 tablespoons) before and after dosing will be done to assess any changes in glucose or insulin. Blood draws will occur at 0, 30, 60, 90, 120, 180, and 240 minutes after dosing.
* Urine samples will be collected throughout the test day to measure the body's response to the daily doses of extract.
* Meet with dietitian to assess food intake to assure it has not changed from normal diet.
* At Day 21 only, a DXA scan will be performed as described above (at Day -3). Females of child-bearing potential will have a urine pregnancy test prior to the DXA scan.

ELIGIBILITY:
Inclusion Criteria:

* Are an overall healthy adult
* Are male or female, ages 18-65 at time of consent
* Are female and of childbearing potential, you must agree to use one of the approved contraception method [(i.e., barrier method, intrauterine and cervical devices, oral contraceptives, hormonal injections (Depo Provera®), condoms with spermicidal gel or foam, contraceptive patch (Ortho Evra), diaphragm, or abstinence)], prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until the follow-up visit.
* Have a BMI within the range 18.5-40 kg/m2 (this is a measure of your height to weight ratio).
* Are capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Have no significant cardiac, pulmonary, gastrointestinal, hepatic, renal, hematological, endocrine, neurological and psychiatric disease
* Have overall normal clinical laboratory tests as deemed by the physician

Exclusion Criteria:

* Have a prior history of Type 1 or 2 diabetes
* Are a female who is pregnant or lactating.
* Are taking certain medications (these will be reviewed with you by the study staff).
* Are anticipating or planning to have surgery during the study period.
* Are a current smoker or have smoked within the previous 6 months.
* Have had a weight change of more than 5% in the last 2 months.
* Are taking prescription or over the counter medications or supplements for weight loss.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Levels of bioactive components from the Russian Tarragon Nutrasorb in the blood and urine | on average weekly for 3 weeks

SECONDARY OUTCOMES:
Glucose tolerance measured with an OGTT | on average weekly for 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer C Rood, Ph.D., Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-26): https://cdn.clinicaltrials.gov/large-docs/03/NCT02088203/Prot_SAP_000.pdf